CLINICAL TRIAL: NCT06090175
Title: The Effect of Using Projector Kaleidoscope and Matching Card on Children's Fear and Physiological Parameters in 3-6 Year Old Children Who Are Administered Inhaler Medication
Brief Title: The Effect of Using Projector Kaleidoscope and Matching Card on Children's Fear and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/14
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-10

CONDITIONS: Fear; Child, Only; Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- projector colleyscope group (Experimental): Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. Before starting the procedure, the child will be introduced to the projector colleidoscope. Before the procedure, this device, which looks like a toy, will be projected onto the wall to divert attention. The projection will continue throughout the inhaler medication administration process. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.
  Interventions: Other: Projector colleyscope group
- Matching card group (Experimental): Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. The child will be allowed to play with the matching cards 2-3 minutes before starting the drug treatment and will then be encouraged to play throughout the procedure. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.
  Interventions: Other: Matching card group
- Control group (No Intervention): Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. Nothing will be shown to the child during the application. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, the Child Fear Scale will be evaluated by the researcher and the parent and recorded by the researcher in the intervention follow-up form.

INTERVENTIONS:
Other: Projector colleyscope group — Projector kaleidoscope will be used in children aged 3-6 who are administered inhaler medication.
  Arms: projector colleyscope group
Other: Matching card group — Matching card will be used in children aged 3-6 who are administered inhaler medication.
  Arms: Matching card group

SUMMARY:
This research was planned as a randomized controlled experimental type to determine the effect of using a projector caleidoscope and matching card on children's fear and physiological parameters in 3-6-year-old children who were administered inhaler medication.

According to the power analysis performed for the sample size, the power of the sample was calculated with the G*Power 3.1 program in line with the literature. While the amount of Type I error was 0.05 and the power of the test was 0.95 (α= 0.05, 1-β= 0.95), the minimal sample size was calculated as 105 children (35 children in each group). Considering the possible losses from the sample for any reason during the study period, it was planned to increase the number of samples by 10% and include 38 children in the study and control groups. The data of the research will be collected using the following data collection tools; Child Information Form and Fear Rating Scale

DETAILED DESCRIPTION:
Discovering ways to reduce/eliminate children's anxiety and fear regarding treatment practices will help children experience less fear and stress during these interventions. Examples of methods that can be used include watching cartoons, blowing up balloons, making bubbles, playing videos or games with virtual reality glasses, listening to music, using a caleidoscope, using distraction cards, clown shows, parents trying to divert attention, and playing toys.

Discovering ways to reduce/eliminate children's anxiety and fear regarding treatment practices will help children experience less fear and stress during these interventions.

This research was planned as a randomized controlled experimental type to determine the effect of using a projector collets-cope and matching card on children's fear and physiological parameters in 3-6-year-old children who were administered inhaler medication.

Place and Time the Research Was Conducted The research will be conducted in Tarsus State Hospital pediatric services. Pediatric 1 ward has 16 beds, the pediatric 2 ward has 20 beds, the infant 2 ward has 20 beds, the infant 1 ward has 16 beds and the pediatric surgery ward has 16 beds. Hospitalizations are made due to bronchitis, tonsillitis, measles, pneumonia, otitis, rheumatoid arthritis, nausea, vomiting, diarrhea, high fever, urinary tract infection, appendicitis, circumcision and scabies.

After obtaining written consent from the parent of the child to be treated with inhaler medication, the parent will be explained about the inhaler medication administration and what will be done during the procedure. Then the descriptive information form will be filled out. Children's physiological parameters (pulse, blood pressure, respiration, SPO2) will be measured before and after the procedure. The parent and nurse will evaluate the child's fear score before and after the procedure, which will be recorded in the follow-up form.

Inhaler drug administration is usually applied 3 times at 20-minute intervals in the clinic. While the first inhaler is being administered, the application will be done with the child sitting, choosing a mask suitable for his/her face. The child should be given an average of 10 minutes. After the inhaler medication is given through the mask for a period of time, the fear score will be evaluated simultaneously by the nurse and the parent.

Projector caleidoscope group: Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. Before starting the procedure, the child will be introduced to the projector caleidoscope. Before the procedure, this device, which looks like a toy, will be projected onto the wall to divert attention. The projection will continue throughout the inhaler medication administration process. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, of the Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.

Matching card group: Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. The child will be allowed to play with the matching cards 2-3 minutes before starting the drug treatment and will then be encouraged to play throughout the procedure. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, of the Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.

Control group: The child was given an average of 10 minutes. Inhaler medication will be provided with a mask that lasts. Nothing will be shown to the child during the application. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, of the Child Fear Scale will be evaluated by the researcher and the parent and recorded by the researcher in the intervention follow-up form.

Data analysis The data obtained within the scope of the research will be evaluated using the Statistical Package For Social Science (SPSS) 26.0 package program. Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of the data. Normal distribution assumptions will be taken into account in the application of hypothesis tests.

Pearson chi-square test will be applied to determine whether the dependent variables are normally distributed according to the groups' characteristics. One Way ANOVA test will be used to compare quantitative continuous data between more than two independent groups. Repeated measurements within the group will be evaluated with the Repeated Measures test. The findings will be evaluated at a 95% confidence interval and a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 3-6 years old,
* No communication problems (visual/auditory/mental),
* Oxygen saturation is 90% or above,
* The child does not have a disease that may affect his/her life,
* Parent and child volunteering to participate in the research.

Exclusion Criteria:

* Nebul drug administration
* The child has a visual, hearing or mental disability

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Child Information Form | 1 day
  The information form was prepared by scanning the literature on the subject and has 12 questions including the child's age, gender, complaint, parent age (who was with him/her during the application) and educational status, physiological parameters before and after inhaler application.
Children's Fear Scale | 1 day
  It is used to evaluate the anxiety/fear level of children. The scale uses cartoon faces consisting of five pictures and the anxiety/fear level is evaluated with numbers between "0" and "4". The first picture shows a score of "0", that is, "no anxiety/fear is felt", and the last picture shows a score of "4", that is, "the most severe anxiety/fear". As the score increases, the level of anxiety/fear also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Korkmaz, Principal Investigator — Tarsus University
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conk, Z. Başbakkal, Z. Yılmaz, H. Bolışık, B. (2013). Pediatri Hemşireliği, Ankara:Akademisyen Tıp Kitabevi.
- [Background] Durak, H. (2019). Çocuklarda İnhaler İlaç Uygulaması Sırasında Çizgi Film İzletme Ve Oyun Kartı Kullanımının Fizyolojik Parametreler ve Korku Düzeyine Etkisi.(Yüksek Lisans Tezi),(645415).
- [Background] Erdinç, E. (2022). Evde Nebülizatör Tedavisi Kime? Nasıl?. Toraks Dergisi, 3(2), 21-25. Retrieved from https://turkthoracj.org/content/files/sayilar/93/buyuk/pdf_Toraksder_197.pdf
- [Background] İnal, S. & Canbulat, N. (2015). Çocuklarda İşlemsel Ağrı Yönetiminde Dikkati Başka Yöne Çekme Yöntemlerinin Kullanımı . Güncel Pediatri , 13 (2) , 116-121
- [Background] Nilsson S, Finnstrom B, Kokinsky E, Enskar K. The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. Eur J Oncol Nurs. 2009 Apr;13(2):102-9. doi: 10.1016/j.ejon.2009.01.003. Epub 2009 Feb 20. PMID 19230769
- [Background] Taşdemir Akkavak, D. & Sarıkaya Karabudak, S. (2019). Hastanede Yatan Okul Çağı Çocukların Hemşireyi ve Hastaneyi Algılama Durumlarının İncelenmesi . Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi , 12 (1) , 46-56
- [Background] Türk Düdükcü, F. & Taş Arslan, F. (2016). Çocuklarda Nebülizatör İle İlaç Uygulama; Problemler Ve Çözüm Önerileri . Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi , 5 (4) , 71-77 .
- [Background] Özsamuri, G. (2020) Maske İle İnhaler İlaç Uygulanan 3-6 Yaş Grubu Çocuklarda Müzik Dinletme Ve Çizgi Film İzletmenin Hissedilen Korku, Anksiyete ve Fizyolojik Parametrelere Etkisinin Belirlenmesi.